CLINICAL TRIAL: NCT02296229
Title: Study of Stereotactic Body Radiotherapy (SBRT) for High-Risk Localized Prostrate Cancer
Brief Title: Stereotactic Body Radiation Therapy in Treating Patients With Localized High-Risk Prostate Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-001427; NCI-2014-02183 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); JCCCID410 (Other: Jonsson Comprehensive Cancer Center); 13-001427 (Other: University of California at Los Angeles Institutional Review Board)
Record Dates: First submitted 2014-11-13; First posted 2014-11-20 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Adenocarcinoma of the Prostate; Stage III Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery; Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (SBRT) (Experimental): Patients undergo SBRT daily or every other day for a total of 5 fraction not exceeding 14 consecutive days. Patients may also receive androgen deprivation therapy for up to 9 months at the discretion of the treating physician.
  Interventions: Radiation: stereotactic body radiation therapy; Other: quality-of-life assessment; Other: laboratory biomarker analysis; Drug: androgen deprivation therapy

INTERVENTIONS:
Radiation: stereotactic body radiation therapy — Undergo SBRT
  Other Names: SBRT; stereotactic radiation therapy; stereotactic radiotherapy
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: laboratory biomarker analysis — Correlative studies
Drug: androgen deprivation therapy — up to 9 months at the discretion of the treating physician
  Other Names: androgen suppression therapy

SUMMARY:
This clinical trial studies stereotactic body radiation therapy in treating patients with high-risk prostate cancer that has not spread to nearby lymph nodes or to other parts of the body. Stereotactic body radiation therapy is a specialized radiation therapy that delivers a single, high dose of radiation directly to the tumor and may kill more tumor cells and cause less damage to normal tissue. Studying quality of life in patients undergoing stereotactic body radiation therapy may help identify the long-term effects of treatment on patients with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the efficacy of stereotactic body radiation therapy (SBRT) in patients with high-risk localized prostate cancer compared to historical data from clinical trials.

II. To establish the safety with physician-reported outcomes after SBRT in patients with high risk localized prostate cancer.

III. To establish the quality of life with patient-reported validated questionnaires after SBRT in patients with high risk localized prostate cancer.

OUTLINE:

Patients undergo SBRT daily or every other day for a total of 5 fraction not exceeding 14 consecutive days. Patients may also receive androgen deprivation therapy for up to 9 months at the discretion of the treating physician.

After completion of study treatment, patients are followed up every 4 months for 1 year, every 6 months for 5 years, and then every 12 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary non-metastatic adenocarcinoma of the prostate
* Risk-group classification into the Dâ€™Amico or National Comprehensive Cancer Network (NCCN) â€˜high-riskâ€™ group, as defined by the presence of any one of the following high-risk factors:

  * Pre-biopsy prostate-specific antigen (PSA) >= 20
  * Biopsy Gleason score 8-10
  * Clinical stage T3
* No pelvic nodal metastases (based on computed tomography [CT] or magnetic resonance imaging [MRI] findings)
* No distant metastases, based upon:

  * CT scan or MRI of the pelvis within 120 days prior to registration
  * Bone scan within 120 days prior to registration; if the bone scan is suspicious, a plain x-ray and/or MRI must be obtained to rule out metastasis
* Karnofsky performance status (KPS) >= 70
* Ability to understand, and willingness to sign, the written informed consent
* Patient will have opted for SBRT among definitive treatment choices

Exclusion Criteria:

* Patients with any evidence of distant metastases
* Hormonal therapy (luteinizing hormone-releasing hormone [LHRH] agonist or oral anti-androgen) exceeding 4 months prior to registration
* Prior cryosurgery, high intensity focused ultrasound (HIFU) or brachytherapy of the prostate
* Prior pelvic radiotherapy
* History of Crohnâ€™s disease or Ulcerative colitis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2014-01-27 (Actual); Primary Completion 2026-01-27 (Estimated); Study Completion 2027-01-27 (Estimated)

PRIMARY OUTCOMES:
Biochemical progression free survival | At 3 years
  Biochemical progression is defined as rising PSA profile of > 2 ng/mL above post-SBRT nadir.
Biochemical progression free survival | At 5 years
  Biochemical progression is defined as rising PSA profile of > 2 ng/mL above post-SBRT nadir.
Incidence of patient-reported genitourinary (GU) and gastrointestinal (GI) toxicity based on the Common Terminology Criteria for Adverse Events (CTCAE) version 4 | At 4 months
Incidence of patient-reported GU and GI toxicity based on the CTCAE version 4 | Up to 5 years
Changes in health related quality of life based on Expanded Prostate Cancer Index Composite questionnaire | Baseline to up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Amar Kishan, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, Los Angeles, California, United States